CLINICAL TRIAL: NCT06201494
Title: Prospective Multicentre Study on Symptoms in First-onset Bronchial Asthma in Children and Adolescents
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jana Tuková, MUDr, Phd, Charles University, Czech Republic
Other Study IDs: CZ-VFN-PEDMET-ASTHMA-001
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Asthma; Asthma in Children; Dyspnea; Cough; Pneumonia; Wheezing; Shortness of Breath; Chest Tightness; Lower Respiratory Tract and Lung Infections; Recurrent Respiratory Tract Infections; Mucus; Plug
MeSH Terms: conditions — Asthma; Dyspnea; Cough; Pneumonia; Respiratory Sounds; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bronchial asthma may present with symptoms other than the commonly reported complaints (cough, chest tightness, shortness of breath and wheezing). Less common symptoms include chronic or recurrent productive cough, inspiratory dyspnoea or recurrent pneumonia. Children presenting with these symptoms are often diagnosed with asthma bronchiale and benefit from antiasthmatic management.

DETAILED DESCRIPTION:
International guidelines for the diagnosis of bronchial asthma list cough, chest tightness, shortness of breath and wheezing as the four basic symptoms of asthma. The diagnosis of bronchial asthma is based on the presence of two or more of these symptoms over time, together with evidence of bronchial hyperresponsiveness and a favourable response to antiasthmatic treatment. In children under 5 years of age, the occurrence of an isolated cough as a possible asthma symptom (cough variant asthma) is also accepted if bronchial hyperresponsiveness is documented and the difficulty subsides on therapy. Pulmonologists also refer children over 5 years of age who have only an isolated cough with no other symptoms before diagnosis.

In practice, however, it is also possible to see children whose asthma initially manifests as conditions assessed as recurrent pneumonia, isolated chronic cough of a moist nature or as inspiratory dyspnoea. These atypical symptoms are not oficially counted as asthma symptoms. In this study, the investigators focus on prevalence of typical and atypical asthma symtpoms. Furthermore, the investigators study sensitivity of offical asthma symptom questinaire ISAAC in children with typical and atypical asthma symptoms.

ELIGIBILITY:
Inclusion Criteria:

- Child 3 - 18 years old, first evaluation in pulmonary outpatient clinic for any of the following respiratory symptoms: cough, shortness of breath, chest tightness, wheezing, recurrent lower respiratory tract and lung infections, dyspnoea of any type, pathological listening findings.

Exclusion Criteria:

* Other documented chronic respiratory, cardiovascular, neurological, genetic, infectious, metabolic disease, significant immaturity or other disease that may be accompanied by respiratory symptoms.

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with suspected diagnosis of asthma without any further chronic disease associated with respiratory symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of typical and atypical asthma symptoms in children with asthma bronchiale | Initial checkup with asthma symptom documentation and answering the ISAAC questionaire. Suspection on asthma diagnosis and initiation of therapy and scheduled follow-up within 3 months to confirm the diagnosis.
  We study prevalence of asthma symptoms in children with newly diagnosed asthma. We monitor atypical and atypical symptoms. Typical symptoms are cough, chest tightness, shortness of breath and wheezing according to current global asthma guidelines (GINA). Atypical symptoms are not yet fully documented in literature but they might be represented by recurrent pneumonia, isolated chronic wet cough or inspiratory dyspnoea. Comparison of sensitivity of ISAAC questionaire in group of children with typical and atypical asthma symptoms. In practice, however, it is also possible to see children whose asthma initially manifests as conditions assessed as recurrent pneumonia, isolated chronic cough of a moist nature or as inspiratory dyspnoea. These atypical symptoms are not oficially counted as asthma symptoms. In our study, we focus on prevalence of typical and atypical asthma symtpoms. We study sensitivity of questionaire ISAAC in children with typical and atypical asthma symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Tukova, MD,PhD, Principal Investigator — Charles University, Czech Republic First Faculty of Medicine, Prague
Locations (1):
- First faculty of Medicine, Charles university., Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available upon publication to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of study and its publication. For 5 years.
Access Criteria: Proposals should be submitted to jana.tukova@vfn.cz.